CLINICAL TRIAL: NCT02915445
Title: T Cells Armed With Chimeric Antigen Receptor Recognizing EpCAM for Patients With Advanced Solid Tumors
Brief Title: EpCAM CAR-T for Treatment of Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Wei Wang, Dr, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKLB-083
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Malignant Neoplasm of Nasopharynx TNM Staging Distant Metastasis (M); Breast Cancer Recurrent; Gastric Cancer With Metastasis
Keywords: EpCAM CAR-T, solid tumors, cancer immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EpCAM CAR-T cells (Experimental): Autologous T cells from patient are engineered to expressing a special chimeric antigen receptor to recognizing EpCAM by lentiviral vector. The engineered T cells were then endowed cytotoxicity to the tumor cells and hold the potential to inhibit the advance of tumors.
  Interventions: Biological: EpCAM CAR-T cells

INTERVENTIONS:
Biological: EpCAM CAR-T cells — Patients included will be infused the autologous T cells armed with CAR recognizing EpCAM. After infusion, cytokines and other medical test will be performed.

SUMMARY:
This study is for patients that have nasopharyngeal carcinoma, breast cancer, gastric cancer and other solid tumors. As epithelial cell adhesion molecule (EpCAM) is a well characterized molecule that is closely with poor prognosis and tumor metastasis and invasion. Many therapies targeting EpCAM have shown benefits for cancer patients. This study is to determine the safety of the engineered T cells armed with chimeric antigen receptor (CAR-T) recognizing EpCAM. At the same time, efficacy is to be evaluated by the criteria of RECIST. The EpCAM CAR-T were produced by lentiviral transduction of the novel 2nd generation of CAR genes. Different cohorts of patients receive EpCAM CAR-T with a dose-escalating manner. This study is to find the largest dose of EpCAM CAR-T, to learn what the adverse effects are and to find out whether this experimental intervention might help patients with nasopharyngeal carcinoma, breast cancer and other EpCAM positive solid tumors.

DETAILED DESCRIPTION:
In this study, the original tumor tissue specimen should be stained to determine the expression levels of EpCAM. Only the patients having tumor with high expression levels will be included.

50-100ml blood with be drawn to get enough CD3 T cells at least 2x10^7. After separation, PBMC will be activated via antibodies of CD3 and CD28 and then transduced by lentivirus bearing the EpCAM CAR gene. Then the EpCAM CAR-T cells will proliferate up to 10-100 folds for infusion. The produced cells will be frozen or infused if available.

Included patients will be preconditioned by cyclophosphamide for lymphodepletion if the levels of white blood cells and lymphocytes are normal. Infusion of T cells, at least 1 day after lymphodepletion, is dose escalating and beginning at the lowest level. If the first level is proven to be safe, the next level will be proceeded. Once severe side effects were observed, the dose will be lowered or the dose will be stopped.

During infusion, patients will be taken care of by cardiogram monitor. Blood drawing will be taken before infusion, at 4h after infusion and on day 4, 7, 14, 30, 60, 90, 120, 150, 180 to determine the presence of CAR-T cells. At the same time, cytokines including IL-6, TNF-alpha and IFN-gamma and C-reactive protein levels will be determined. Routine imaging studies will be proceeded.

To see whether there are long-term side effects of this therapy, patients received CAR-T cells will be followed up to at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at the time of procurement:

* Recurrent or refractory nasopharyngeal carcinoma and breast cancer and other solid tumors.
* Karnofsky score of greater than or equal to 60.
* Informed consent explained to, understood by and signed by subject/guardian. -
* Subject/guardian given copy of informed consent

Treatment Inclusion criteria:

* Recurrent or refractory EpCAM-positive nasopharyngeal carcinoma, breast cancer, gastric cancer and other epithelial tumors determined by Immunohistochemistry (IHC) or RT-PCR. EpCAM expression in tumors on IHC should be greater than or equal to grade 2 and greater than or equal to 2+ intensity score. Wherein grades are defines as: Grade 0: no staining; Grade 1: 1-25%; Grade 2: 26-50% and Grade 3: 51-100% of cell staining for EpCAM and intensity scores are: negative; 1+; 2+ and 3+ using breast cancer standard arrays as a guide for intensity.
* Age ≥ 18 years
* Life expectancy ≥ 6 weeks
* Karnofsky score ≥ 60
* Bilirubin less than or equal to 3x normal, AST less than or equal to 5x normal,
* ALT less than or equal to 5x, serum creatinine less than or equal to 2x upper limit of normal for age, and Hgb greater than or equal to 8.0
* Pulse oximetry of greater than or equal to 90% on room air.
* Sexually active subjects must be willing to utilize one of the more effective birth control methods for 6 months after the T cell infusion. The male partner should use a condom.
* Available autologous transduced T lymphocytes with greater than or equal to 20% expression of EpCAM CAR determined by flow-cytometry and killing of EpCAM-positive targets greater than or equal to 20% in cytotoxicity assay.
* Subjects should have been off other investigational antineoplastic therapy for two weeks prior to entry in this study.
* Cyclophosphamide will be allowed 72 hours preinfusion.
* Dexamethasone up to a total dose of 2 mg per day will be allowed if medically indicated.
* Informed consent explained to, understood by and signed by research subjects/guardian.
* Subject/guardian given copy of informed consent.

Exclusion Criteria:

Exclusion Criteria at the time of procurement:

* Known HIV positivity.

Treatment Exclusion Criteria:

* Severe intercurrent infection.
* Known HIV positivity.
* Pregnant or lactating.
* History of hypersensitivity reactions to murine protein-containing products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events/dose limiting toxicity as assessed by CTCAE v4.0 | 6 weeks after infusion
  Determine the largest dose of EpCAM CAR-T cells for patients with nasopharyngeal carcinoma, breast cancer and other tumors expressing EpCAM.

SECONDARY OUTCOMES:
Response rate of participants treated with EpCAM CAR-T cells assessed by RECIST v1.1 | 24 months after infusion of the CAR-T cells
  Determine whether there is therapeutic efficacies of the safe dose infusion of EpCAM CAR-T cells for patients with solid tumors.
Persistence of EpCAM CAR-T cells and correlation with the Response rate | 24 months post CAR-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Ph.D, Principal Investigator — State Key Laboratory of Biotherapy, Cancer Center, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osta WA, Chen Y, Mikhitarian K, Mitas M, Salem M, Hannun YA, Cole DJ, Gillanders WE. EpCAM is overexpressed in breast cancer and is a potential target for breast cancer gene therapy. Cancer Res. 2004 Aug 15;64(16):5818-24. doi: 10.1158/0008-5472.CAN-04-0754. PMID 15313925
- [Background] Burges A, Wimberger P, Kumper C, Gorbounova V, Sommer H, Schmalfeldt B, Pfisterer J, Lichinitser M, Makhson A, Moiseyenko V, Lahr A, Schulze E, Jager M, Strohlein MA, Heiss MM, Gottwald T, Lindhofer H, Kimmig R. Effective relief of malignant ascites in patients with advanced ovarian cancer by a trifunctional anti-EpCAM x anti-CD3 antibody: a phase I/II study. Clin Cancer Res. 2007 Jul 1;13(13):3899-905. doi: 10.1158/1078-0432.CCR-06-2769. PMID 17606723
- [Background] Stoecklein NH, Siegmund A, Scheunemann P, Luebke AM, Erbersdobler A, Verde PE, Eisenberger CF, Peiper M, Rehders A, Esch JS, Knoefel WT, Hosch SB. Ep-CAM expression in squamous cell carcinoma of the esophagus: a potential therapeutic target and prognostic marker. BMC Cancer. 2006 Jun 23;6:165. doi: 10.1186/1471-2407-6-165. PMID 16796747
- [Background] Spizzo G, Went P, Dirnhofer S, Obrist P, Moch H, Baeuerle PA, Mueller-Holzner E, Marth C, Gastl G, Zeimet AG. Overexpression of epithelial cell adhesion molecule (Ep-CAM) is an independent prognostic marker for reduced survival of patients with epithelial ovarian cancer. Gynecol Oncol. 2006 Nov;103(2):483-8. doi: 10.1016/j.ygyno.2006.03.035. Epub 2006 May 6. PMID 16678891
- [Background] Murakami N, Mori T, Yoshimoto S, Ito Y, Kobayashi K, Ken H, Kitaguchi M, Sekii S, Takahashi K, Yoshio K, Inaba K, Morota M, Sumi M, Itami J. Expression of EpCAM and prognosis in early-stage glottic cancer treated by radiotherapy. Laryngoscope. 2014 Nov;124(11):E431-6. doi: 10.1002/lary.24839. Epub 2014 Jul 14. PMID 25043563
- [Background] Deng Z, Wu Y, Ma W, Zhang S, Zhang YQ. Adoptive T-cell therapy of prostate cancer targeting the cancer stem cell antigen EpCAM. BMC Immunol. 2015 Jan 31;16(1):1. doi: 10.1186/s12865-014-0064-x. PMID 25636521